CLINICAL TRIAL: NCT07245875
Title: Analysis of the Safety and Efficacy of Administering Umbilical Cord Mesenchymal Stem Cell Secretome in Patients With Severe Erectile Dysfunction Non-responsive to Sildenafil
Brief Title: Umbilical Cord Mesenchymal Stem Cell Secretome Administration in Severe Erectile Dysfunction Non-responsive to Sildenafil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Ria Margiana, M.D., Ph.D, Indonesia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-04-0512; PUTI Q1 (Other: Universitas Indonesia)
Record Dates: First submitted 2025-08-03; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Erectile Dysfunction; Diabetes Mellitus Type 2
Keywords: erectile dysfunction; non responsive to sildenafil; secretome; Umbilical Cord Mesenchymal Stem Cell
MeSH Terms: conditions — Erectile Dysfunction; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- severe erectile dysfunction non responsive to Sildenafil (Experimental)
  Interventions: Biological: Intracavernosal Injection of Umbilical Cord Mesenchymal Stem Cell Secretome

INTERVENTIONS:
Biological: Intracavernosal Injection of Umbilical Cord Mesenchymal Stem Cell Secretome — UC-MSC secretome was obtained from UC-MSC cultures with 80% confluence in serum-free medium after 24 hours of incubation The VEGF level in the secretome given was 1400 pg/ml.
  The intervention was the administration of 0.5 mL/site of secretome injection injected intra-cavernous to all subjects using a 22-gauge needle according to a sterile protocol. The same volume was given at bilateral sites of the penile shaft. The intra-cavernous injection sites were in the right and left dorsolateral regions of the penis. After the intervention, tolerability was assessed by observing and questioning the subjects regarding pain during injection.

SUMMARY:
The study is an experimental pre-post-test design involving 12 patients with severe ED non-responsive to sildenafil. Safety parameters included pain, hematoma, local bleeding, and infection, while efficacy was measured using the IIEF-5 questionnaire, EHS, and morning erection.

DETAILED DESCRIPTION:
The study employed umbilical cord mesenchymal stem cell secretome, one intravenous injection containing one ml into two locations, one injection in one cavernous body, and three direct follow-ups with the patient: directly after injection, one day and one month after the injection.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 40-65 years who undergo treatment at the Andrology Clinic of RSUD Dr. Soetomo.
* Severe erectile dysfunction caused by organic factors for at least 6 months, based on an IIEF-5 score of 5-7
* History of undergoing treatment with sildenafil 100 mg for four sessions.
* Evaluation of IIEF-5 score < 22 and not meeting the MCID criteria, defined as an IIEF-5 score increase of less than 4
* Type II Diabetes Melitus with an HbA1c test result of < 7%.
* Laboratory test results for liver function (SGOT and SGPT) and kidney function (urea and creatinine) are within normal limits.
* Patients with undergoing treatment with antidepressant.

Exclusion Criteria:

* Anatomical abnormalities of the penis that are clinically visible, such as Peyronie's disease, a history of priapism, a history of penile implants, skin irritation, and lesions in the area surrounding the penile skin.
* Active and significant systemic or local infection.
* History of bleeding or blood clotting disorder therapy.
* History of systemic autoimmune disorders and immunosuppressive treatment
* History of prostate surgery, history of malignancy, or a PSA level > 4 ng/mL.
* Untreated hypogonadism or low serum total testosterone (<200 ng/dL).
* Uncontrolled hypertension or hypotension (systolic blood pressure >170 or <90 mmHg, and diastolic blood pressure >100 or <50 mmHg).
* Unstable cardiovascular disease (e.g., unstable angina, myocardial infarction within the last 6 months, and congestive heart failure).

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients with severe erectile dysfunction non-responsive sildenafil
Enrollment: 12 (Actual)
Dates: Start 2024-04-12 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | one day and one month
  A visual analog is used for measuring pain. The patient will be asked to describe the pain on scale 1 to 10. Scale 1 means no pain and 10 means very great pain. A higher score indicates a worse outcome.
Hematomes | one day and one month
  Hematomes means blue discoloration. 0 scale means ther is no discoloration and 1 means there is discoloration.
Bleeding | one day and one month
  Bleeding is one of the outcomes of the research. If there is bleeding, it would be marked as 1; if there is no bleeding, it would be marked as 0.
Erection Hardness Score | One month
  Rapid diagnostic tool to evaluate erectile dysfunction. There are 4 scores. 1 indicate severe erectile dysfunction (worst) and 4 indicates there is optimal erection (good).
IIEF-5 | One month
  Rapid diagnostic tool to evaluate erectile dysfunction
Restrictive Index | one month
PSV | one month
SPL | one month
FPL | one month
Penile Circumference | one month

CONTACTS AND LOCATIONS:
Locations (1):
- Univesitas Indonesia Hospital, Depok, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2025-10-06): https://cdn.clinicaltrials.gov/large-docs/75/NCT07245875/Prot_000.pdf
  • Statistical Analysis Plan (2025-10-06): https://cdn.clinicaltrials.gov/large-docs/75/NCT07245875/SAP_001.pdf
  • Informed Consent Form (2025-10-06): https://cdn.clinicaltrials.gov/large-docs/75/NCT07245875/ICF_002.pdf